CLINICAL TRIAL: NCT03814915
Title: DIabetes REsearCh on Patient straTification
Acronym: DIRECT
Status: Completed | Type: Observational
Sponsor: Lund University (Other)
Responsible Party: Sponsor
Other Study IDs: IMIDIRECT_2012
Record Dates: First submitted 2019-01-21; First posted 2019-01-24 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Type2 Diabetes
Keywords: Gene-environment interaction; Genome; Glycaemic control; Lifestyle; Microbiome; Prediabetes; Proteome; Type 2 diabetes
MeSH Terms: conditions — Prediabetic State; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood Omics: Fasting blood samples taken for genomic, transcriptomic, proteomic and metabolomic assessments.
  Microbiome Urine Toenail clippings
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study 1 - Prediabetes: The primary objective of Study 1 is to collect biosamples and information that might yield novel, predictive biomarkers for glycaemic deterioration in non-diabetic high-risk participants.
  Participants in Study 1 were recruited from existing prospective cohort studies in or around each of the following European cities: Malmö, Sweden (Malmö Diet and Cancer Study); Amsterdam, The Netherlands (Hoorn Study); Copenhagen, Denmark (Inter99); and Kuopio, Finland (METSIM). A clinically practicable screening tool (DIRECT-DETECT) was used to identify at-risk participants from existing cohort studies, who were then recruited into this new prospective cohort study (Study 1).
- Study 2- Diabetic: The primary objective of Study 2 is to collect biosamples and information that might yield novel, predictive biomarkers for glycaemic deterioration in people who have recently been diagnosed with type 2 diabetes. Participants in Study 2 of DIRECT are recruited from or nearby each of the following European cities: Malmö, Sweden; Amsterdam, the Netherlands; Copenhagen, Denmark; Exeter, UK; Newcastle, UK; Dundee, UK. Potential participants are recruited through targeted searches of existing databases and research registers combined with person-to-person contact at educational clinics and through routine retinal screening programmes.

SUMMARY:
The overarching goal of the IMI DIRECT (Innovative Medicines Initiative Diabetes Research on Patient Stratification) Consortium is the identification of biomarkers that aid therapeutic targeting in prediabetes (Study 1) or early onset type 2 diabetes (Study 2).

DETAILED DESCRIPTION:
There are two multicentre prospective cohort studies within the glycaemic deterioration work package of IMI DIRECT (WP2). These two cohorts are designed to address the area of glycaemic deterioration by amassing data and biomaterials that will be used to discover novel biomarkers for glycaemic deterioration in people at high risk of developing type 2 diabetes (Study 1) and in those who have recently been diagnosed with the disease (Study 2).

ELIGIBILITY:
Study 1

Inclusion criteria

* No treatment with insulin-sensitising, glucose-lowering or other antidiabetic drugs
* Fasting capillary blood glucose <10 mmol/l at baseline
* White European (self-report of parental ethnicity)
* Age ≥35 and <75 years

Exclusion criteria

* Diagnosed diabetes of any type, HbA1c ≥6.5% (48 mmol/mol) or fasting plasma glucose ≥7.0 mmol/l or 2 h plasma glucose >11.0 mmol/l previously
* For women, pregnancy, lactation or plans to conceive within the study period
* Use of a pacemaker
* Any other significant medical reason for exclusion as determined by the investigator

Study 2

Inclusion Criteria:

* Patients diagnosed with type 2 diabetes not less than 6 months and not more than 24 months before baseline examination
* Management by lifestyle with or without metformin therapy
* All HbA1c <7.6% (<60 mmol/mol) within previous 3 months
* White European
* Age ≥35 and <75
* Estimated GFR >50 ml/min'

Exclusion Criteria:

* Type 1 diabetes

  * A previous HbA1c >9.0% (>75 mmol/mol)
  * Prior treatment with insulin or an oral hypoglycaemic agent other than metformin
  * BMI <20 or >50 kg/m2
  * Pregnancy, lactation or plans to conceive within the study period
  * Any other significant medical reason for exclusion as determined by the investigator

Ages: 35 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: White European (self-report of parental ethnicity), Age ≥35 and <75 years
Sampling Method: Probability Sample
Enrollment: 3049 (Actual)
Dates: Start 2012-10-15 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Glycemic deterioration | Up to 10 years follow-up
  Change in glucose (or HbA1c) over time and/or progression to anti diabetic medications/insulin

CONTACTS AND LOCATIONS:
Overall Officials: Ewan Pearson, FRCP, Principal Investigator — University of Dundee; Paul W Franks, PhD, Principal Investigator — Lund University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Koivula RW, Heggie A, Barnett A, Cederberg H, Hansen TH, Koopman AD, Ridderstrale M, Rutters F, Vestergaard H, Gupta R, Herrgard S, Heymans MW, Perry MH, Rauh S, Siloaho M, Teare HJ, Thorand B, Bell J, Brunak S, Frost G, Jablonka B, Mari A, McDonald TJ, Dekker JM, Hansen T, Hattersley A, Laakso M, Pedersen O, Koivisto V, Ruetten H, Walker M, Pearson E, Franks PW; DIRECT Consortium. Discovery of biomarkers for glycaemic deterioration before and after the onset of type 2 diabetes: rationale and design of the epidemiological studies within the IMI DIRECT Consortium. Diabetologia. 2014 Jun;57(6):1132-42. doi: 10.1007/s00125-014-3216-x. Epub 2014 Apr 4. PMID 24695864
- [Derived] Lyu L, Fan Y, Vogt JK, Clos-Garcia M, Bonnefond A, Pedersen HK, Dutta A, Koivula R, Sharma S, Allin KH, Brorsson C, Cederberg H, Chabanova E, De Masi F, Dermitzakis E, Elders PJ, Blom MT, Hollander M, Eriksen R, Forgie I, Frost G, Giordano GN, Grallert H, Haid M, Hansen TH, Jablonka B, Kokkola T, Mahajan A, Mari A, McDonald TJ, Musholt PB, Pavo I, Prehn C, Ridderstrale M, Ruetten H, Hart LM', Schwenk JM, Stankevic E, Thomsen HS, Vangipurapu J, Vestergaard H, Vinuela A, Walker M, Hansen T, Linneberg A, Nielsen HB, Brunak S, McCarthy MI, Froguel P, Adamski J, Franks PW, Laakso M, Beulens JWJ, Pearson E, Pedersen O. The dynamics of the gut microbiota in prediabetes during a four-year follow-up among European patients-an IMI-DIRECT prospective study. Genome Med. 2025 Jul 15;17(1):78. doi: 10.1186/s13073-025-01508-7. PMID 40665409
- [Derived] Atabaki-Pasdar N, Ohlsson M, Vinuela A, Frau F, Pomares-Millan H, Haid M, Jones AG, Thomas EL, Koivula RW, Kurbasic A, Mutie PM, Fitipaldi H, Fernandez J, Dawed AY, Giordano GN, Forgie IM, McDonald TJ, Rutters F, Cederberg H, Chabanova E, Dale M, Masi F, Thomas CE, Allin KH, Hansen TH, Heggie A, Hong MG, Elders PJM, Kennedy G, Kokkola T, Pedersen HK, Mahajan A, McEvoy D, Pattou F, Raverdy V, Haussler RS, Sharma S, Thomsen HS, Vangipurapu J, Vestergaard H, 't Hart LM, Adamski J, Musholt PB, Brage S, Brunak S, Dermitzakis E, Frost G, Hansen T, Laakso M, Pedersen O, Ridderstrale M, Ruetten H, Hattersley AT, Walker M, Beulens JWJ, Mari A, Schwenk JM, Gupta R, McCarthy MI, Pearson ER, Bell JD, Pavo I, Franks PW. Predicting and elucidating the etiology of fatty liver disease: A machine learning modeling and validation study in the IMI DIRECT cohorts. PLoS Med. 2020 Jun 19;17(6):e1003149. doi: 10.1371/journal.pmed.1003149. eCollection 2020 Jun. PMID 32559194